CLINICAL TRIAL: NCT05188027
Title: Acute Glycemic Effects of Aerobic and Resistance Exercise in Post-menopausal Women With Type 1 Diabetes
Brief Title: Aerobic vs Resistance Exercise in Post-menopausal Women With Type 1 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Women and Children's Health Research Institute, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00107673
Record Dates: First submitted 2021-12-08; First posted 2022-01-12 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Type 1 Diabetes; Post-menopause
Keywords: Exercise; Physical activity
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity | interventions — Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): All participants will take part in all three testing conditions
  Interventions: Other: Aerobic Exercise; Other: Resistance Exercise; Other: No exercise

INTERVENTIONS:
Other: Aerobic Exercise — Walking at 60% of maximal aerobic capacity on a treadmill
Other: Resistance Exercise — Performing one set of 10 repetitions of 10 different weight-lifting exercises
Other: No exercise — Participants will rest in a supine position for 30 minutes.

SUMMARY:
Participants will be asked to wear a continuous glucose monitor for at least three days on three separate occasions. One testing session will be a no-exercise resting control session (90 minutes). One will be a moderate aerobic exercise session (30 minutes of exercise, 60 minutes of recovery), and the third will be a moderate weight-lifting session (~30 minutes of exercise, 60 minutes of recovery).The investigators will measure changes in blood glucose during exercise by drawing blood during and after exercise. Post-exercise glucose trends will be examined using continuous glucose monitoring.

DETAILED DESCRIPTION:
Pre-test measures: Interested participants will be invited to either the Exercise Physiology laboratory the Augustana campus of the University of Alberta, or the Physical Activity and Diabetes Laboratory on the main campus of the University of Alberta. They will be asked questions related to menopause, PA levels, and medication. Blood pressure and heart rate will also be measured. Where participants are eligible, anthropometric characteristics will be measured using standard protocols. A blood sample will be drawn for assessment of HbA1c. Those who meet all eligibility criteria and complete informed consent forms will be asked to complete the initial exercise tests. Participants will perform a maximal aerobic capacity test with ECG monitoring, under the supervision of a certified exercise physiologist. Indirect calorimetry will be used to assess oxygen consumption and carbon dioxide production and will be used to extrapolate the participant's aerobic capacity. Participants will undergo a strength test for each of the ten exercises involved in the study, in order to estimate the their 1 repetition maximum. Participants will also be asked to undergo a dual energy x-ray absorptiometry (DXA) scan for body composition in the Clinical Research Unit at the Alberta Diabetes Institute. While this procedure generally requires proof of a negative pregnancy test, participants will be provided with a waiver in order to decline this test (in light of their menopausal status).

Testing sessions: Participants will be asked to arrive at the lab at around 4:00 pm for all three sessions, which will be randomly assigned. During the sessions, participants will be asked to perform one of the three activities: 1) seated rest 2) aerobic exercise (walking on a treadmill at 50% of the participant's pre-determined VO2max) or 3) resistance exercise consisting of 1 set of 10 repetitions of 10 different exercises with 90 seconds rest between sets. Blood samples will be drawn at baseline, after 10, 20 and 30 minutes of exercise, along with 30- and 60-minutes post-exercise via an IV catheter. Indirect calorimetry will be used to ensure that the participant is exercising at the appropriate intensity. Participants will be asked to match their daily food and insulin intake as closely as possible from one testing session to the next for the day before, day of and day after the testing session. The investigators will provide them with log sheets to assist in this task. They will also be asked to avoid strenuous exercise and alcohol intake.

A CGM sensor will be subcutaneously inserted by one of the investigators (trained by a group from the CGM manufacturer) into the anterior abdominal area of the participant, or on the back of the arm of the participant, approximately 2 days prior to the first testing session. The Dexcom G6 CGM receiver will store glucose data every 5 minutes for up to 10 days. The participant will be instructed on how to remove their sensor at least 24 hours after the exercise session, and will be asked to return the receiver to enable the upload of their data to Dexcom Clarity by the study team.

Interviews: During the third and final testing session, study participants will be invited to answer questions about their study participation experience, exercise preferences, barriers to exercise, and other information they feel may improve their exercise experience. These interviews will be audio recorded and transcribed.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes, diagnosed for at least one year
* post-menopause (at least one year since last menstrual period), or have had a hysterectomy and bilateral salpingo oophorectomy
* able to perform aerobic and resistance exercise
* able to visit the lab in Edmonton, Alberta (University of Alberta)

Exclusion Criteria:

* HbA1c > 9.9 %
* frequent and unpredictable hypoglycemia
* change in insulin management strategy within the last 2 months
* blood pressure > 140 / 95
* severe peripheral neuropathy
* history of cardiovascular disease
* musculoskeletal injuries interfering with exercise performance
* use of medications (other than insulin) that affect glucose metabolism
* BMI > 30 kg/m2
* smoking
* moderate to high alcohol intake (> 2 drinks/day)

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Blood glucose | From 0 minutes to 45 minutes (beginning to the end of exercise/control) and then for 60 minutes after exercise
  Change in blood glucose

SECONDARY OUTCOMES:
mean continuous glucose monitoring (CGM) glucose | 6 hours, 12 hours, nocturnal (midnight to 6am) and 24 hours post-exercise
  mean of all measurements over the selected time frames
coefficient of variation (CV) of CGM glucose | 6 hours, 12 hours, nocturnal (midnight to 6am) and 24 hours post-exercise
  CV of CGM glucose over the selected time frames
standard deviation (SD) | 6 hours, 12 hours, nocturnal (midnight to 6am) and 24 hours post-exercise
  SD of CGM glucose over the selected time frames
frequency of hypoglycemia | 6 hours, 12 hours, nocturnal (midnight to 6am) and 24 hours post-exercise
  number of times that CGM glucose is equal to or less than 3.9 mmol/L
frequency of hyperglycemia | 6 hours, 12 hours, nocturnal (midnight to 6am) and 24 hours post-exercise
  number of times that CGM glucose is equal to or greater than 10.0 mmol/L
percent time spent in hyperglycemia | 6 hours, 12 hours, nocturnal (midnight to 6am) and 24 hours post-exercise
  percentage of time spent with CGM glucose equal to or greater than 10.0 mmol/L
percent time spent in hypoglycemia | 6 hours, 12 hours, nocturnal (midnight to 6am) and 24 hours post-exercise
  percentage of time spent with CGM glucose equal to or lower than 3.9 mmol/L
percent time spent in range | 6 hours, 12 hours, nocturnal (midnight to 6am) and 24 hours post-exercise
  percent of time spent with CGM glucose between 4.0 and 9.9 mmol/L
carbohydrate supplementation | from 0 minutes to 45 minutes (during exercise)
  grams of carbohydrate provided during exercise to prevent hypoglycemia

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Alberta Diabetes Institute, Edmonton, Alberta
  - Institut de recherches cliniques de Montréal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No